CLINICAL TRIAL: NCT01245452
Title: Comparative Study of the Clinical Response and Cardiorespiratory Endurance in Early Rheumatoid Arthritis Patients Treated With Tocilizumab or Methotrexate Addendum Protocol : Global Gene Expression Profiles in Synovial Biopsies
Brief Title: Study of the Response and Cardiorespiratory Endurance in Early RA Patients Treated With Tocilizumab or Methotrexate
Acronym: TOMERA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Patrick Durez (Other)
Responsible Party: Sponsor-Investigator, Patrick Durez, Professeur clinique, Université Catholique de Louvain
Organization: Université Catholique de Louvain (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P1200/002
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Tocilizumab; Cardiorespiratory endurance
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tocilizumab (Experimental): Tocilizumab (8 mg/kg monthly from week 0 to 20)
  Interventions: Drug: Tocilizumab
- Methotrexate (Active Comparator): MTX at a dose ranging from 10 mg/week at baseline to 20 mg/week at week 8
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab (8 mg/kg monthly from week 0 to 20)
  Other Names: Roche EU/1/08/492/001; ATC code L04AC07
  Arms: Tocilizumab
Drug: Methotrexate — MTX at a dose ranging from 10 mg/week at baseline to 20 mg/week at week 8
  Arms: Methotrexate

SUMMARY:
To measure the CRE by a work capacity index obtained in a submaximal testing (W65%/kg) in early RA patients treated with tocilizumab compared to Methotrexate alone.

The secondary endpoints : analyze the clinical efficacy of Tocilizumab in this population and correlate the CRE response with other marker (CRP, Hb, DAS, HAQ) and evaluate the safety profile of Tocilizumab.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is the most prevalent (about 1%) inflammatory rheumatic disorder.

Interleukin-6 (IL-6) has emerged as a potential therapeutic target in RA. This is based on the greater understanding of the role this cytokine can play in various aspects of the pathogenesis of RA. It has been shown that IL-6 is responsible for various clinical symptoms, including,fatigue, anemia, anorexia, fever, as well as the production of autoantibodies and increase in the erythrocyte sedimentation rate, all of which develop in patients with RA. Tocilizumab, as monotherapy and in combination with methotrexate, has been shown to be effective for RA patients with insufficient response to methotrexate or other disease-modifying antirheumatic drugs. These observations about the effects of tocilizumab were extended to patients refractory to tumor necrosis factor inhibitors. Tocilizumab also slows down the progression of structural joint damage. Furthermore, a 5-year long-term safety and efficacy has been shown. The place of Tocilizumab therapy in early RA is still unknown.

Cardiorespiratory endurance (CRE), the most fundamental component of physical fitness can be severely impaired in patients with rheumatoid arthritis (RA). It has been shown that intensive and early treatment of RA can induce sustained clinical remission, improve general health and physical fitness and might therefore have an impact on the quality of life of RA patient. This study was planned to measure the CRE by a work capacity index obtained in a submaximal testing (W65%/kg) in early RA patients treated with tocilizumab compared to Methotrexate alone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA (according to American College of Rheumatology ACR criteria)
* Disease duration < 2 years.
* Age between 18 and 70 years old.
* Active RA defined by a disease activity score 28 DAS28-CRP score > 3.2 with a swollen joint count ≥ 4
* MTX naive
* Stable therapy with corticosteroids or nonsteroidal anti-inflammatory drug NSAIDs
* Presence of knee arthralgia or synovitis (addendum protocol with synovial biopsy).

Exclusion Criteria:

Previous MTX treatment. Exclusion for severe physical handicap to perform CRE. Exclusion for general safety (history of severe allergic reaction, sepsis, malignancy within 5 years, pregnancy, severe heart failure) Concurrent treatment with other DMARDs than MTX or any anti-TNF and biological therapies.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To measure the CRE by a work capacity index obtained in a submaximal testing (W65%/kg) in early RA patients treated with tocilizumab compared to Methotrexate alone. | 2 years
  not necessary

SECONDARY OUTCOMES:
To analyze the clinical efficacy of Tocilizumab in this population. | 2 years
  no necessary
To correlate the CRE response with other marker (CRP, Hb, Disease activity score DAS, HAQ). | 2 years
  no necessary
To evaluate the safety profile of Tocilizumab. | 2 years
  no necessary
To assess the effect of Tocilizumab on synovial histopathology of early RA | 2 years
  not necessary

CONTACTS AND LOCATIONS:
Overall Officials: Patrick DUREZ, Md, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Université Catholique de Louvain, Brussels, Belgium